CLINICAL TRIAL: NCT02129907
Title: The Purpose of the Study is to Examine Whether Iron Deficiency Anemia is Associated With Increased Production of Thrombin and Whether Correction of Anemia by Providing Iron Intravenously Causes a Significant Reduction in Production of Thrombin.
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Elias mazen, prof mazen elias, HaEmek Medical Center, Israel
Other Study IDs: thrombingeneration- anemia
Record Dates: First submitted 2014-05-01; First posted 2014-05-02 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2015-12

CONDITIONS: Iron Deficiency Anemias
Keywords: Anemias; Iron-Deficiency; thrombin
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Weeks
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In total 50 subjects with iron deficiency anemia treated with intravenous iron are planned for inclusion in this trial. After signing an informed consent a blood sample will be obtained from each participant before iron treatment. The investigators will measure the thrombin generation in plasma assessed by the calibrated automated thrombogram (CAT). patient will go face to face interview and will be asked to answer structured questionnaire which will include information on demographics, clinical data ( fever, allergies , etc.) and comorbidities

Two weeks after completing intravenous iron administration additional blood samples will be taken: thrombin generation will be measured

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* Iron deficiency anemia that did not response to oral iron treatment and is planned to receive iron supplement intravenously.
* Signing the informed consent

exclusion criteria:

* chronic inflammatory disease
* renal failure
* Malignancy
* Infectious disease
* Other reason for anemia except iron deficiency anemia.
* Pregnant women
* Use of anti aggregating agents or anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men and women over age 18 suffering from iron deficiency anemia that wasnt responded to oral iron treatment or there is contraindication for oral iron therapy.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
thrombin generation levels | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek medical center, Afula, Israel